CLINICAL TRIAL: NCT06049550
Title: The Influence of the Thickening of Bowman's Capsule on the Clinical Prognosis of Patients With Diabetic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2023-0174
Record Dates: First submitted 2023-09-07; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Kidney Disease; Extracellular Matrix Alteration
Keywords: Diabetic Kidney Disease; extracellular matrix; parietal epithelial cells
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild thicknening of Bowman's Capsule
  Interventions: Other: no intervention
- severe thickening of Bowman's Capsule
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Diabetic kidney disease (DKD) is the leading cause for renal replacement therapy in developed country. DKD is also the primary cause of ESKD among middle-aged and elderly people in China. Renal pathological markers have been proved to have clinical and prognostic value in both non diabetic and diabetic kidney diseases. To discriminate lesions by various degrees of severity, the Working Group of the Renal Pathology Society (RPS) developed a pathologic classification for DKD in 2010. The classification is based on glomerular lesions, with a separate evaluation for interstitial and vascular lesions. In a decade, there were several new characteristics common to DKD, such as the presence of mesangiolysis, glomerular hyalinosis, segmental sclerosis and extracapillary hypercellularity, which have been noted in patients with diabetes and may have prognostic importance. But it is still unclear whether thickening of Bowman's capsule predicts the progression of DKD.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥ 18 years old, male or female 2) Patients diagnosed as diabetes kidney disease by renal biopsy

Exclusion Criteria:

* 1) Patients combined with non diabetes kidney disease; 2) Patients with kidney transplant failure; 3) Patients undergoing zero point puncture for kidney transplantation; 4) less than 5 glomeruli in the renal puncture sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosised as diabetic kidney disease by renal biopsy from January 1, 2017 to December 31, 2021 in Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, the First Affiliated Hospital of China Medical University, Shanghai Sixth People's Hospital and Shanghai General Hospital.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
renal failure | From the diagnosis of diabetes kidney disease by renal biopsy to December 31, 2022
  estimated glomerular filtration rate（eGFR）<15ml/min/1.73m2, renal replacement treatment or death caused by renal disease

IPD SHARING:
Plan to Share IPD: Undecided